CLINICAL TRIAL: NCT04647838
Title: A Phase II Study of Tepotinib in Patients With Solid Cancers Harboring c-MET Amplification or Exon 14 Mutation Who Progressed After Standard Treatment for Advanced/Metastatic Disease
Brief Title: Tepotinib in Solid Tumors Harboring MET Alterations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chungbuk National University Hospital (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KM08
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Solid Tumor; MET Exon 14 Skipping Mutation; MET Amplification
Keywords: solid tumors; MET Exon 14; MET Amplification; cMET; lung; neoplasm; cMET amplification; METex14; cancer; MET Exon 14 skipping
MeSH Terms: conditions — Neoplasms | interventions — tepotinib; EMD1214063

STUDY DESIGN:
Intervention Model Description: Experimental: Arm 1_NSCLC Patients with non-small cell lung cancer (NSCLC) harboring MET alteration Experimental: Arm 2_Other solid tumors Solid tumors excluding NSCLC harboring MET alteration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NSCLC (Experimental): Tepotinib 500mg (2 tablets of 250mg) per day D1-21 orally, once daily
  Interventions: Drug: Tepotinib
- Other cancers (Experimental): Tepotinib 500mg (2 tablets of 250mg) per day D1-21 orally, once daily
  Interventions: Drug: Tepotinib

INTERVENTIONS:
Drug: Tepotinib — Tepotinib 500mg (2 tablets of 250mg) per day D1-21 orally, once daily
  Other Names: MSC2156119J; EMD 1214063

SUMMARY:
The aim of this study is to understand efficacy of tepotinib in patients with solid cancers harbouring c-MET amplification or exon 14 mutation who progressed after standard treatment for metastatic disease.

DETAILED DESCRIPTION:
This study is a basket trial with two strata(NSCLC and other cancer). If MET exon 14 skipping mutation or MET amplification(copy number gain ≥6.0 ) is detected by NGS method, then confirmation of genetic findings by Molecular Steering Committee will be followed. Patient can participate in this trial after confirmation of genetic analysis and reviewing other inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed solid cancers (NSCLC, gastric cancer, colorectal cancer, breast cancer, hepatocellular cancer, head and neck cancer, RCC and other solid cancers)
2. Subjects who are not eligible for surgical and/or local-regional therapies or who have progressive disease (PD) after surgical and/or local-regional therapies
3. Subjects who have disease progression or are intolerant to the prior standard treatment for advanced solid cancers
4. A tumor biopsy (excluding fine needle aspiration and cytology samples) is required for determining MET status (a fresh pretreatment tumor biopsy is recommended but archived tumor sample is acceptable).
5. Patients with MET exon 14 skipping mutation detected by NGS method and c-MET copy number gain (≥6.0) in the archival or fresh tumor tissue specimen identified in K-MASTER panel. All genetic findings must be reviewed by the study Molecular Steering Committee, prior to study entry.
6. Male or female, 19 years of age or older
7. Measurable disease in accordance with Response Evaluation Criteria in Solid Tumors (RECIST v 1.1). The target lesion that has received previous local therapy should not be considered as measurable unless clear progression has been documented since the therapy.
8. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
9. Signed and dated informed consent indicating that the subject has been informed of all the pertinent aspects of the trial prior to enrollment
10. Life expectancy judged by the Investigator of at least 3 months

Exclusion Criteria:

1. Eligibility criteria:

1. Histologically or cytologically confirmed solid cancers (NSCLC, gastric cancer, colorectal cancer, breast cancer, hepatocellular cancer, head and neck cancer, RCC and other solid cancers)
2. Subjects who are not eligible for surgical and/or local-regional therapies or who have progressive disease (PD) after surgical and/or local-regional therapies
3. Subjects who have disease progression or are intolerant to the prior standard treatment for advanced solid cancers
4. A tumor biopsy (excluding fine needle aspiration and cytology samples) is required for determining MET status (a fresh pretreatment tumor biopsy is recommended but archived tumor sample is acceptable).
5. Patients with MET exon 14 skipping mutation detected by NGS method and c-MET copy number gain (≥6.0) in the archival or fresh tumor tissue specimen identified in K-MASTER panel. All genetic findings must be reviewed by the study Molecular Steering Committee, prior to study entry.
6. Male or female, 19 years of age or older
7. Measurable disease in accordance with Response Evaluation Criteria in Solid Tumors (RECIST v 1.1). The target lesion that has received previous local therapy should not be considered as measurable unless clear progression has been documented since the therapy.
8. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
9. Signed and dated informed consent indicating that the subject has been informed of all the pertinent aspects of the trial prior to enrollment
10. Life expectancy judged by the Investigator of at least 3 months

2. Exclusion criteria

1. Prior treatment with any agent targeting the HGF/c-MET pathway
2. Prior EGFR therapy for EGFR activating mutant NSCLC
3. Patients who received local treatment within 4 weeks prior to the first administration of tepotinib (e.g., major surgery, radiation therapy, hepatic arterial embolization, transcatheter arterial chemoembolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation). NOTE: palliative radiotherapy should be completed at least 7 days prior to the first administration of the tepotinib.
4. Prior history of organ transplant
5. Laboratory index at screening(refer to protocol)
6. Past or current history of neoplasm other than current cancer, except for curatively treated non-melanoma skin cancer, in situ carcinoma of the cervix, node-negative thyroid cancer or other cancer curatively treated and with no evidence of disease for at least 3 years
7. Known central nervous system (CNS) or brain metastasis that is either symptomatic or untreated
8. Medical history of difficulty swallowing, malabsorption, or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested products
9. Clinically significant gastrointestinal bleeding within 4 weeks prior to the first administration of tepotinib.
10. Impaired cardiac function(refer to protocol)
11. Hypertension uncontrolled by standard therapies (not stabilized to ≤ 150/90 mmHg)
12. Subject with a family history of long QT syndrome or who take any agent that is known to prolong QT/QTc interval or with a marked prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval > 450 msec)
13. Known human immunodeficiency virus (HIV) infection
14. Subjects who were diagnosed with acute pancreatitis and/or chronic pancreatitis by related symptoms or imaging study.
15. Known or suspected drug hypersensitivity to any ingredients of tepotinib
16. Female subjects who are pregnant or lactating, or males and females of reproductive potential not willing or not able to employ a highly effective method of birth control/contraception to prevent pregnancy from 2 weeks before receiving study drug until 3 months after receiving the last dose of study drug. A highly effective method of contraception is defined as having a low failure rate (< 1% per year) when used consistently and correctly.
17. Concurrent treatment with anti-cancer therapy
18. Substance abuse, other acute or chronic medical or psychiatric condition that may increase the risk associated with trial participation in the opinion of the Investigator
19. Participation in another interventional clinical trial within 28 days prior to the first administration of tepotinib or within a time period that is less than the cycle length for the investigational treatment (whichever is shorter), or if the subject has any AE caused by the investigational treatment that has not recovered to Grade 0-1
20. Previous anticancer treatment-related toxicities not recovered to baseline or Grade 1 (except alopecia) prior to administratin of tepotinib
21. Subjects with any concurrent medical condition or disease that will potentially compromise the conduct of the study at the discretion of the Investigators
22. Clinically significant third space fluid accumulation (despite the use of diuretics), e.g., uncontrolled pleural effusion or ascites
23. Uncontrolled venous or arterial thromboembolism

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rates (RECIST1.1) | Baseline up to 20 months
  Objective response will be determined according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by investigator.
  Objective response is defined as either a confirmed complete response (CR) or partial response (PR) from first administration of trial treatment to first observation of progressive disease (PD). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in the sum of the longest diameter (SLD) of all lesions. PD is defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.

SECONDARY OUTCOMES:
Progression free survival | Baseline until PD or death within 84 days of last tumor assessment; assessed up to 20 months
  Progression free survival as assessed by investigators is defined as the time (in months) from the first administration of trial treatment to the date of the first documentation of PD (based on independent review) or death due to any cause within 84 days of the last tumor assessment, whichever occurs first
Disease control rate | Baseline up to 20 months
  Objective disease control is defined as either a confirmed CR or PR, or stable disease (SD) lasting at least 12 weeks (84 days) as assessed by investigator. CR: Disappearance of all evidence of target and non-target lesions.
Overall survival | Baseline until death, assessed up to 20 months
  Overall survival is defined as the time (in months) from first trial treatment administration to the date of death.
Toxicity and drug compliance | From the first dose of study drug administration until 33 days after the last dose of study drug administration, assessed up to 20 Months
  This outcome measure will be presented as the percentage of subjects with any adverse event (AE). Percentages are calculated using total number of subjects per treatment cohort as the denominator.

CONTACTS AND LOCATIONS:
Overall Officials: Ki Hyeong Lee, M.D., Study Chair — Chungbuk National University Hospital
Locations (22):
- South Korea (22):
  - Chonnam National University Hwasun Hospital, Hwasun, Chonnam
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Dankook University Hospital, Cheonan
  - Keimyung University Dongsan Hospital, Daegu
  - Konyang University Hospital, Daejeon
  - National Cancer Center, Goyang-si
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - Gachon University Gil Medical Center, Incheon
  - The Catholic University of Korea Incheon St. Marry Hospital, Incheon
  - Gyeongsang National University Hospital, Jinju
  - Inje University Haeundae Pain Hospital, Pusan
  - Kosin University Gaspel Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam-si
  - Chungang University Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No